CLINICAL TRIAL: NCT00919061
Title: A Phase II Study of Gemcitabine and Cisplatin Plus Sorafenib in Patients With Advanced Biliary Tract Carcinomas Naïve to Systemic Therapy
Brief Title: Gemcitabine and Cisplatin Plus Sorafenib in Patients With Advanced Biliary Tract Carcinomas Naive to Systemic Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-029
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer
Keywords: GALL BLADDER; BILE DUCTS; BAY 43-9006; SORAFENIB; CISPLATIN; GEMCITABINE; 09-029
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Gemcitabine; Cisplatin; Sorafenib

ARMS (1):
- Gemcitabine and Cisplatin plus Sorafenib (Experimental): This is a non-randomized, open label, single institution, phase II study of gemcitabine and cisplatin plus sorafenib for the treatment of patients with advanced or biliary tract carcinomas naïve to systemic therapy.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Sorafenib

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine: 800 mg/m^2 over 30 minutes IV, weekly for 2 weeks, followed by a week off treatment.
Drug: Cisplatin — 20 mg /m^2 over 30 minutes IV, weekly for 2 weeks, followed by a week off treatment.
Drug: Sorafenib — 400 mg PO once a day continuously.

SUMMARY:
The purpose of this study is to test an investigational combination of drugs for bile duct or gallbladder cancers.

Gemcitabine and cisplatin are two forms of chemotherapy commonly used in combination to treat bile duct and gallbladder cancers. We are looking to improve treatment results. We will attempt to do so by adding sorafenib (a type of monoclonal antibody) to your treatment plan. Sorafenib acts by attaching to blocking specific targets on cells. These targets may help the cancer cells grow and divide. This study will help answer the question of whether sorafenib is a helpful drug in patients with bile duct or gallbladder cancers when given with gemcitabine and cisplatin.

This study is a phase 2 study. The purpose of a phase 2 study is to find out what effects, good and/or bad, sorafenib in combination with gemcitabine and cisplatin has on advanced bile duct and gallbladder cancers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically / cytologically verified, non-resectable, recurrent, or metastatic biliary tract carcinoma including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma and gallbladder carcinoma. Combined cholangiocarcinoma and hepatocellular carcinoma is allowed.Patients must have uni-dimensionally measurable disease by x-ray, CT scan, MRI scan or physical examination.
* KPS ≥ 80%
* Age ≥ 18 years
* Adequate bone marrow function defined as: Hb ≥ 8 g/dl, ANC ≥ 1.5 K/mcL, Platelets ≥ 100 K/mcL
* Adequate renal function defined as Serum creatinine < 2.0 mg/dl and calculated creatinine clearance ≥ 60 ml/min using the formula:
* Cockcroft-Gault formula:

Cockcroft-Gault Formula - MALES CrCl = (140 - age[years]) (body wt[kg]) (72) (serum creatinine [mg/dL]) Cockcroft-Gault Formula - FEMALES CrCl = 0.85 x male value

* If calculated creatinine clearance is not within range using the above formula, then measured levels from 24-hour urine collection may be used to calculate the creatinine clearance.
* Adequate hepatic function defined as total bilirubin ≤ 2 mg/dl, ALT/AST/ ≤ 3 x ULN (≤ 5 if liver metastases). Patients with biliary obstruction can join if bilirubin corrects to required limit after adequate biliary drainage.
* PT/INR ≤ 1.7 and PTT ≤ 1.5 x ULN, unless the patient is receiving anti-coagulation therapy with agents such as warfarin or heparin
* Patients who have received prior local therapy, i.e. embolization, radiation therapy, etc. (except for chemoembolization) are eligible provided that measurable disease falls outside the treatment field or within the field but has shown an increase of ≥20% in the size. Prior local therapy must be completed at least 4 weeks prior to the baseline scan
* Women of childbearing potential must have a negative pregnancy test.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter. Patients are encouraged to continue barrier method contraception for two years or longer after treatment.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Any previous chemotherapy, biologic therapy, or investigational agent, except for 5-FU or gemcitabine given as adjuvant therapy as single agents and/or as radio-sensitizing agents. Patient must have completed adjuvant therapy no less than six months prior to accrual. Patients with previous significant allergic hypersensitivity to gemcitabine are excluded.
* Evidence of another active cancer that may influence patient outcome as determined by the Principal Investigator, except for non-melanoma skin carcinoma, melanoma in-situ, in-situ carcinoma of the cervix curatively treated, treated superficial bladder cancer, and adenocarcinoma of the prostate that has been surgically treated with a post-treatment PSA that is non-detectable.
* Known brain metastases
* History of primary central nervous system tumors or brain metastases, and/or seizures not well controlled with standard medical therapy.
* Uncontrolled intercurrent illness including, but not limited to psychiatric illness/social situations that would limit compliance with study requirements.
* Known HIV positive patient
* Blood Pressure of > 150/100 mm Hg
* Significant cardiovascular disease including congestive heart failure (New York Heart Association Class II or higher) or active angina pectoris.
* History of a myocardial infarction within 6 months.
* History of a stroke or transient ischemic attack within 6 months.
* Clinically significant peripheral vascular disease.
* Evidence of bleeding diathesis or coagulopathy.
* Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks.
* Uncontrolled infection.
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.
* Pregnant (positive pregnancy test)
* Breast-feeding should be discontinued if the mother is to be treated on clinical trial.
* Serious non-healing wound, ulcer, or bone fracture
* Use of St. John's Wort or rifampin (rifampicin)
* Any condition that impairs patient's ability to swallow whole pills
* Any malabsorption problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ghassan Abou-Alfa, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine and Cisplatin Plus Sorafenib: This is a non-randomized, open label, single institution, phase II study of gemcitabine and cisplatin plus sorafenib for the treatment of patients with advanced or biliary tract carcinomas naïve to systemic therapy.
  Gemcitabine and Cisplatin plus Sorafenib: Patients will receive treatment under the following schedule:
  Gemcitabine: 800 mg/m2 over 30 minutes IV, weekly for 2 weeks, followed by a week off treatment.
  Cisplatin: 20 mg /m2 over 30 minutes IV, weekly for 2 weeks, followed by a week off treatment.
  Sorafenib: 400 mg PO once a day continuously. Three weeks of treatment correspond to one cycle.
Period: Overall Study
Arm/Group | Gemcitabine and Cisplatin Plus Sorafenib
Started | 39
Completed | 37
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine and Cisplatin Plus Sorafenib
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Progression free survival will be calculated from study entry to documented disease progression, death from any cause, or drop out due to toxicity, whichever occurs first.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine and Cisplatin Plus Sorafenib
Number analyzed (Participants) | 37
percentage of participants | 51 [34 to 66]

2. Primary Outcome: Median PFS
Description: as for outcome 1
Time Frame: 6 mos
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine and Cisplatin Plus Sorafenib
Number analyzed (Participants) | 37
months
  Progression Free Survival | 6.5 [3.5 to 8.3]
  Overall Survival | 14.4 [11.6 to 19.2]

ADVERSE EVENTS:
Arm/Group | Gemcitabine and Cisplatin Plus Sorafenib
Serious Adverse Events (participants affected / at risk) | 24/39
Other Adverse Events (participants affected / at risk) | 37/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine and Cisplatin Plus Sorafenib (N=39)
Ascites (Gastrointestinal disorders) | 2 (2)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (2)
Blood disorder (Investigations) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1)
Colitis, infectious (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Death-Disease Progression (General disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Fever (General disorders) | 5 (6)
Fistula, GU - Vagina (Reproductive system and breast disorders) | 1 (1)
Gastrointestinal, other (Gastrointestinal disorders) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Hemorrhage/Bleeding, other (Blood and lymphatic system disorders) | 1 (1)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 2 (2)
Infection (Infections and infestations) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3)
Neutrophil count decreased (Investigations) | 2 (2)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain-Other (General disorders) | 3 (3)
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Platelet count decrease (Investigations) | 3 (3)
Renal failure (Renal and urinary disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Thrombosis (Vascular disorders) | 8 (9)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Vision-blurred vision (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine and Cisplatin Plus Sorafenib (N=39)
Alanine aminotransferase increased (Investigations) | 11 (30)
Aspartate aminotransferase increased (Investigations) | 8 (12)
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 (59)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 16 (69)
Serum amylase increased (Investigations) | 8 (26)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Blood bilirubin increased (Investigations) | 6 (19)
Constipation (Gastrointestinal disorders) | 5 (5)
Creatinine increased (Investigations) | 2 (13)
Diarrhea (Gastrointestinal disorders) | 6 (10)
Fatigue (General disorders) | 17 (25)
Hyperglycemia (Metabolism and nutrition disorders) | 17 (68)
Anemia (Blood and lymphatic system disorders) | 30 (366)
Hypertension (Vascular disorders) | 2 (2)
Infection, other (Infections and infestations) | 3 (3)
White blood cell decreased (Investigations) | 16 (66)
Lipase increased (Investigations) | 13 (24)
Lymphocyte count decreased (Investigations) | 9 (15)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (5)
Neutrophil count decreased (Investigations) | 15 (64)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Chest pain (General disorders) | 2 (2)
Pain-other (General disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (20)
Platelet count decreased (Investigations) | 16 (35)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (8)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Rash-Hand Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 10 (13)
Hyponatremia (Metabolism and nutrition disorders) | 4 (11)
Thrombosis (Vascular disorders) | 5 (5)
Tinnitus (Ear and labyrinth disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes